CLINICAL TRIAL: NCT04768166
Title: Phase 2 Pharmacological Trial to Evaluate the Safety of Miglustat Administration in Subjects With Spastic Paraplegia 11 (TreatSPG11)
Brief Title: Testing Miglustat Administration in Subjects With Spastic Paraplegia 11
Acronym: TreatSPG11
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS Fondazione Stella Maris (Other)
Responsible Party: Principal Investigator, Filippo Maria Santorelli, Director Molecular Medicine, Neurogenetics and Neuromuscular Disorders, IRCCS Fondazione Stella Maris
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TreatSPG11; 2019-002827-14 (EudraCT Number)
Record Dates: First submitted 2021-02-12; First posted 2021-02-24 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Hereditary Spastic Paraparesis
Keywords: Autophagic Lysosome Reformation; SPG11; Miglustat; Lisosomal Storage Disorders
MeSH Terms: conditions — Spastic Paraplegia, Hereditary | interventions — miglustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluate the safety of Miglustat administration in subjects with Spastic Paraplegia 11 (Experimental): 100 mg of Miglustat, 3 caps per day for first 4 weeks; 100 mg of Miglustat, 6 caps per day for 8 weeks
  Interventions: Drug: Miglustat 100 MG

INTERVENTIONS:
Drug: Miglustat 100 MG — 100mg/TID in 4w then 200mg/TID in 8 w
  Other Names: Genorph

SUMMARY:
Hereditary spastic paraparesis type 11 (SPG11) is caused by mutations in the SPG11 gene that produces spatacsin, a protein involved in lysosomal function. Studies performed in skin cells (fibroblasts) from SPG11 patients, mice and zebrafish models of the disease showed that the material accumulated in the lysosomes is made of glycosphingolipids (GSL).

Miglustat is a drug that inhibits an enzyme called glucosylceramide synthetase (GCS) which is used for the production of GSL. Miglustat, therefore, helps to delay the production of GSL. This study aims to collect preliminary data on the safety of miglustat on the SPG11 disease and to assess biomarkers.

DETAILED DESCRIPTION:
We will analyze the safety of Miglustat

ELIGIBILITY:
Inclusion Criteria:

* Written signed informed consent;
* Confirmed diagnosis of SPG11;
* Age > 13 years;
* SPRS score ≥ 10 or ≤35;
* Use of effective contraceptive methods and the performance of pregnancy tests (only fertile subjects).

Exclusion Criteria:

* Diagnosis of other concomitant neurodegenerative diseases;
* Outcomes of severe pre- or peri-natal suffering;
* Age ≤ 13 years;
* SPRS score ≥ 35 or ≤10;
* Hypersensitivity or intolerance to miglustat;
* Participation in other pharmacological studies within 30 days of the first Study visit (T0);
* The inability to take the drug;
* Any additional medical conditions;
* Subjects with severe renal impairment;
* Refusal to use effective contraceptive methods and the performance of pregnancy tests (only fertile subjects).

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
1-Changes from baseline blood tests at 24 weeks 2-Changes from baseline neurophysiological tests at 24 weeks 3-Report of severe adverse events | At baseline, 24 weeks
  routine blood test

SECONDARY OUTCOMES:
Changes from baseline GM2/GM3 levels at 24 weeks | At baseline, 24 weeks
  lipid assessments
Assess changes in the scores of the Spastic Paraplegia Rating Scale (SPRS) at 24 weeks | At baseline, 24 weeks
  SPRS rates disease severity (0-52) with lower numbers indicating less impairement

CONTACTS AND LOCATIONS:
Overall Officials: Filippo M Santorelli, MD PhD, Principal Investigator — IRCCS Stella Maris
Locations (1):
- IRCCS Fondazione Stella Maris, Pisa, PI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bellofatto M, De Michele G, Iovino A, Filla A, Santorelli FM. Management of Hereditary Spastic Paraplegia: A Systematic Review of the Literature. Front Neurol. 2019 Jan 22;10:3. doi: 10.3389/fneur.2019.00003. eCollection 2019. PMID 30723448
- [Background] Boutry M, Branchu J, Lustremant C, Pujol C, Pernelle J, Matusiak R, Seyer A, Poirel M, Chu-Van E, Pierga A, Dobrenis K, Puech JP, Caillaud C, Durr A, Brice A, Colsch B, Mochel F, El Hachimi KH, Stevanin G, Darios F. Inhibition of Lysosome Membrane Recycling Causes Accumulation of Gangliosides that Contribute to Neurodegeneration. Cell Rep. 2018 Jun 26;23(13):3813-3826. doi: 10.1016/j.celrep.2018.05.098. PMID 29949766
- [Background] Branchu J, Boutry M, Sourd L, Depp M, Leone C, Corriger A, Vallucci M, Esteves T, Matusiak R, Dumont M, Muriel MP, Santorelli FM, Brice A, El Hachimi KH, Stevanin G, Darios F. Loss of spatacsin function alters lysosomal lipid clearance leading to upper and lower motor neuron degeneration. Neurobiol Dis. 2017 Jun;102:21-37. doi: 10.1016/j.nbd.2017.02.007. Epub 2017 Feb 22. PMID 28237315
- [Background] Lo Giudice T, Lombardi F, Santorelli FM, Kawarai T, Orlacchio A. Hereditary spastic paraplegia: clinical-genetic characteristics and evolving molecular mechanisms. Exp Neurol. 2014 Nov;261:518-39. doi: 10.1016/j.expneurol.2014.06.011. Epub 2014 Jun 20. PMID 24954637
- [Background] Platt FM, Jeyakumar M, Andersson U, Heare T, Dwek RA, Butters TD. Substrate reduction therapy in mouse models of the glycosphingolipidoses. Philos Trans R Soc Lond B Biol Sci. 2003 May 29;358(1433):947-54. doi: 10.1098/rstb.2003.1279. PMID 12803928